CLINICAL TRIAL: NCT00796458
Title: Phase III Study of Chemo-hormonal Therapy Versus Hormonal Therapy Alone in Advanced Hormone-naives Prostate Cancer Patients.
Brief Title: Androgen Ablation With or Without Docetaxel in Treating Patients With Advanced Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O.U. San Giovanni Battista di Torino, Italy (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GOUP-01/04; CDR0000626194 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT 2004-003495-11; EU-20892
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-11

CONDITIONS: Pain; Prostate Cancer
Keywords: pain; adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Pain; Prostatic Neoplasms | interventions — Docetaxel

ARMS (2):
- Arm I (Active Comparator): Patients continue to receive LHRH-A therapy until disease progression.
  Interventions: Drug: releasing hormone agonist therapy
- Arm II (Experimental): Patients receive LHRH-A therapy as in arm I. Patients also receive docetaxel IV on day 1. Treatment with docetaxel repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: releasing hormone agonist therapy

INTERVENTIONS:
Drug: docetaxel — Given IV
  Arms: Arm II
Drug: releasing hormone agonist therapy — Patients receive luteinizing hormone-releasing hormone analogue therapy until disease progression.

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Androgen ablation therapy may lessen the amount of androgens made by the body. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving androgen ablation therapy together with docetaxel is more effective than giving androgen ablation therapy alone in treating patients with advanced prostate cancer.

PURPOSE: This randomized phase III trial is studying androgen ablation and docetaxel to see how well they work compared with androgen ablation alone in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the 2-year progression-free survival rate (biological progression and/or clinical progression) in patients with advanced prostate cancer treated with androgen ablation with vs without docetaxel.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the time to treatment failure in patients treated with these regimens.
* Compare the toxicity profiles of these regimens in these patients.
* Compare the PSA response rate in patients treated with these regimens.
* Compare the response rate in patients with measurable disease treated with these regimens.
* Compare the percentage of patients who undergo PSA normalization.
* Compare the quality of life of patients treated with these regimens.
* Compare the efficacy of these regimens in controlling bone pain in these patients.
* Compare the changes in chromogranin A levels in patients treated with these regimens.
* Compare the total cost of care of patients treated with these regimens.

OUTLINE: This is a multicenter study.

Patients receive luteinizing hormone-releasing hormone analogue (LHRH-A) therapy for 6 months. Patients also receive antiandrogen therapy during the first 5 weeks of LHRH-A therapy. After 6 months of LHRH-A therapy, patients with PSA response are randomized to 1 of 2 treatment arms.

* Arm I: Patients continue to receive LHRH-A therapy until disease progression.
* Arm II:Patients receive LHRH-A therapy as in arm I. Patients also receive docetaxel IV on day 1. Treatment with docetaxel repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients complete questionnaires during treatment to assess bone pain. Quality of life is also assessed.

After completion to study therapy, patients are followed for ≥ 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Meets one of the following criteria

  * Metastatic disease
  * Systemic progressive disease after locoregional therapy (surgery or radiotherapy)
  * No metastatic disease AND meets one of the following criteria:

    * Circulating PSA levels ≥ 50 ng/mL (confirmed by ≥ 2 subsequent evaluations)
    * Biochemical progression with a PSA doubling time < 6 months (with ≥ 3 measurements taken 1 month apart) after primary locoregional treatment (radical prostatectomy or radiotherapy) with curative intent
    * Prostate-confined tumor with high-risk features whose therapy of choice is androgen deprivation
* No symptomatic brain metastases or leptomeningeal disease

PATIENT CHARACTERISTICS:

* ECOG or Zubrod performance status 0-2
* Life expectancy ≥ 6 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 2.0 mg/dL
* AST/ALT ≤ 1.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* No active infection requiring IV antibiotics
* No active ulcer, unstable diabetes mellitus, or other contraindication to corticotherapy
* None of the following cardiovascular conditions:

  * Uncompensated heart failure (ejection fraction < 40%)
  * Myocardial infarction or revascularization procedure within the past 6 months
  * Unstable angina pectoris
  * Uncontrolled cardiac arrhythmia
* No other severe clinical condition that, in the judgment of the local investigator, would place the patient at undue risk or interfere with the study
* Not a prisoner
* No prior malignancy, except for non-melanoma skin cancer, in situ cervical carcinoma, or other cancer that was curatively treated with no evidence of disease for ≥ 5 years
* No familial, social, or geographical condition or significant neurologic or psychiatric disorder that would preclude understanding or rendering informed consent or fully complying with study treatment and follow-up

PRIOR CONCURRENT THERAPY:

* At least 5 years since prior radiotherapy outside the prostate
* Prior hormonal therapy allowed provided it was administered for ≤ 6 months
* At least 12 months since prior hormonal therapy
* More than 30 days since prior participation in another clinical trial involving investigational agents
* No prior surgical castration
* Concurrent androgen deprivation for prostate cancer allowed provided it was started ≤ 3 months prior to initiation of study treatment
* Concurrent anticoagulant treatment allowed
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-04; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate

SECONDARY OUTCOMES:
Overall survival
Time to treatment failure
Toxicity as assessed by NCI CTCAE criteria
PSA response rate (> 50% reduction from baseline)
Disease response rate as assessed by RECIST criteria (in patients with measurable disease)
PSA normalization (normal range 0-4 ng/mL)
Quality of life
Efficacy of treatment in controlling bone pain
Changes in chromogranin A levels
Cost analysis

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Bertetto, MD, Principal Investigator — Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino; Isabella Chiappino, MD — A.O.U. San Giovanni Battista di Torino, Italy
Locations (1):
- Rete Oncologica Piemontese - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin, Italy